CLINICAL TRIAL: NCT06835543
Title: Assessment of Amnion Membrane Versus Chorion Membrane for Soft Tissue Healing After Tooth Extraction; a Randomized Clinical Trial
Brief Title: Soft Tissue Healing After Tooth Extraction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: soft tissue healing
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Badly Broken Maxillary Premolars Indicated for Extraction; Badly Broken Down Vital Teeth
Keywords: Amnion membrane; chorion membrane; soft tissue healing; tooth extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: blinding of outcome assessors and participants will be achieved as the different outcomes will be assessed for all groups by assessors other than the researchers doing the procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amnion membrane (Active Comparator): the amnion membrane tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material
  Interventions: Procedure: Amnion membrane.
- Chorion membrane. (Active Comparator): chorion membrane (Bioxclude , Snoasis Medical , USA) tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material.
  Interventions: Procedure: Chorion membrane

INTERVENTIONS:
Procedure: Amnion membrane. — the amnion membrane tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 5-0 resorbable suture material
  Arms: Amnion membrane
Procedure: Chorion membrane — chorion membrane tucked over the extraction socket then the socket plug will be maintained in place with approximating sutures using 4-0 resorbable suture material.
  Arms: Chorion membrane.

SUMMARY:
Statement of the problem: Tooth extraction results in hard and soft tissue loss which complicates prosthodontic rehabilitation, So different techniques of alveolar ridge preservation should be done to maintain hard and soft tissue dimensions.

Aim: The aim of this study is to compare the effect of amnion membrane versus chorion membrane on soft tissue healing among socket preservation procedure.

DETAILED DESCRIPTION:
Aim: The aim of this study is to compare the effect of amnion membrane versus chorion membrane on soft tissue healing among socket preservation procedure.

Materials and Methods: This parallel arm, randomized controlled clinical trial will involve systemically free patients with remaining roots or badly decayed teeth in the posterior region not indicated for immediate implant placement. They will be randomly allocated to two equal groups. Group A (n=95) socket will be grafted with HAM particulate and the socket will be covered with amnion membrane, and group B (n=95) socket will be grafted with HAM particulate and the socket will be covered with chorion membrane. Soft tissue healing will be assessed (1ry outcome) every day for the first week, day after day second week, once in third and fourth week. Postoperative pain and swelling will be recorded daily by the patient for the 1st two weeks post surgically. Postoperative medication will be prescribed to the patient and postoperative instructions will be explained in detail. Follow-up will be performed to assess the parameters and to ensure performing proper oral hygiene. Data collected will be tabulated and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need simple extraction not indicated for immediate implant placement.

Exclusion Criteria:

1. Patients with inability or anticipated failure to maintain adequate oral hygiene.
2. Pregnant or breast-feeding mothers.
3. Any medical condition or therapy that can affect healing.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Soft tissue healing | every day for the first week, day after day second week, once in third and fourth week
  Surface area/intraoral scanner

SECONDARY OUTCOMES:
Healing index | every day for the first week, day after day second week, once in third and fourth week
  Score (from o to 10, were 0 is no healing and 10 complete healing of tissue )

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of oral and dental medicine , Suez university, Suez, Suez Governorate, Egypt